CLINICAL TRIAL: NCT03656380
Title: A Multi-center, Randomized, Double Blind, Parallel-arm, Placebo Controlled Trial of Mepolizumab for Treatment of Adults and Adolescents With Active Eosinophilic Esophagitis and Dysphagia-predominant Symptoms
Brief Title: Mepo for Eosinophilic Esophagitis (EoE) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: GlaxoSmithKline (Industry); University of Utah (Other); Northwestern University (Other); MNGI Digestive Health, P.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-0431
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: EoE; Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — mepolizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mepolizumab 300 mg (Experimental): Subjects will receive Mepolizumab 300 mg subcutaneously (SQ) monthly for 6 months
  Interventions: Drug: Mepolizumab 300 mg
- Placebo, followed by Mepolizumab 100 mg (Other): This arm will receive placebo, followed by Mepolizumab 100 mg. Subjects will receive placebo subcutaneously (SQ) monthly for 3 months, followed by Mepolizumab 100 mg subcutaneously (SQ) monthly for 3 months. Mepolizumab will be administered with 2 SQ injections of placebo and 1 SQ injection of Mepolizumab 100 mg to maintain blinding.
  Interventions: Drug: Mepolizumab 100 mg; Other: Placebo

INTERVENTIONS:
Drug: Mepolizumab 300 mg — Mepolizumab 300 mg subcutaneous injection
  Other Names: Nucala
  Arms: Mepolizumab 300 mg
Drug: Mepolizumab 100 mg — Mepolizumab 100 mg subcutaneous injection
  Other Names: Nucala
  Arms: Placebo, followed by Mepolizumab 100 mg
Other: Placebo — Saline subcutaneous injection
  Other Names: Saline
  Arms: Placebo, followed by Mepolizumab 100 mg

SUMMARY:
Multi-center, randomized, double blind, parallel-arm, placebo controlled trial to determine whether mepolizumab is more effective than placebo for improving symptoms of dysphagia and decreasing esophageal eosinophil counts in adults and adolescents with active eosinophilic esophagitis (EoE) after an initial 3 month treatment course, and will also assess the impact of an additional 3 months of treatment.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double blind, parallel-arm, placebo controlled trial of mepolizumab. After the first 3 month blinded phase, there will be a second 3 month blinded phase where all patients receive active medication, but the dose will be lower in the subjects initially randomized to the placebo arm.

In the first arm, subjects will receive mepolizumab 300 mg SQ monthly for 3 months. In the second arm, subjects will receive a placebo SQ injection monthly for 3 months. Both groups will have the injection administered under direct observation in a Clinical & Translational Research Center (CTRC) or other clinic to ensure proper administration and compliance. Each visit will also provide an opportunity for symptom questionnaires to be completed and for blood samples to be drawn. After 3 months (the time point where the primary outcome is assessed), all subjects initially randomized to active treatment will continue with mepolizumab dosing 300 mg SQ monthly, and will remain blinded. All subjects initially randomized to placebo will receive mepolizumab 100mg SQ monthly, and will remain blinded. Of note, no dietary changes, changes in baseline Proton Pump Inhibitor (PPI) medication dose, changes in inhaled or intranasal steroid doses, or administration or oral, topical/swallowed, or systemic steroids will be allowed during the study period. Subjects will undergo endoscopy after the first blinded phase (at 3 months) and after the second blinded phase (after 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Age 16-75
* Diagnosis of EoE (eosinophilic esophagitis) as per consensus guidelines (including PPI non-response)*
* Active eosinophilia on esophageal biopsy, with a peak count of least 15 EOS/hpf (eosinophils per high power field) from at least one esophageal level.
* Biopsies from the stomach and duodenum that have ruled out alternative etiologies in all children and in adults with abnormal endoscopic findings or when other gastric or small intestinal conditions are clinical possibilities. If these samples have been obtained during a previous endoscopic evaluation and in the judgement of the site-Investigator the patient has not had a clinically significant change that would merit repeat gastric/duodenal biopsies, then prior normal gastric and duodenal biopsies are acceptable to exclude alternate etiologies.
* Active symptoms of dysphagia with more than 3 episodes of dysphagia over a period of 2 weeks during the screening period, and an Eosinophilic Esophagitis Symptom Activity Index (EEsAI; see below for details) score of ≥ 27 at baseline.
* Able to read, comprehend, and sign consent form.
* Have maintained a stable diet for 6 weeks prior to enrollment.
* Able to maintain a stable diet throughout the duration of the study period.
* Female subjects of childbearing potential who have had their first menses agree to use a highly effective method of birth control during the study and for 30 days after the last dose of study drug. Female subjects with reproductive potential who are using systemic contraceptives (e.g., oral contraceptives, injectable contraceptives, implantable/insertable hormonal contraceptive products, or transdermal patches) to prevent pregnancy must have stable use for ≥28 days prior to screening.

  * PPI non-response is defined as >15 eos/hpf after at least 6 weeks of high dose administration (40mg total per day or higher) of any approved PPI medication or documented evidence of intolerance or allergy to PPIs. The length of the PPI trial period or documented intolerance/allergy will be determined according to the local clinical standard of care.

Exclusion Criteria:

* Esophageal dilation within 8 weeks of the screening endoscopy.
* Inability to pass a standard upper endoscope (8-10mm) due to esophageal narrowing or stricturing.
* Swallowed/topical steroids for EoE within 4 weeks of the screening endoscopy, or a course of systemic corticosteroids within 8 weeks of the screening endoscopy.
* Not having maintained a stable diet for at least 6 weeks preceding the screening endoscopy.
* Initiation, discontinuation, or change of dose regimen of PPIs; leukotriene inhibitors; or nasal, inhaled, and/or orally administered topical corticosteroids for any condition (such as gastroesophageal reflux disease, asthma, or allergic rhinitis) within the 8 weeks prior to the qualifying esophagogastroduodenoscopy (EGD).
* Presence of concomitant eosinophilic gastritis (EG), eosinophilic gastroenteritis (EGE), eosinophilic colitis (EC), Crohn's disease, ulcerative colitis, or celiac disease.
* History of malignancy within 5 years prior to screening, except completely treated in situ carcinoma of the cervix and completely treated non-metastatic squamous or basal cell carcinoma of the skin.
* History of achalasia.
* Prior esophageal surgery.
* History of bleeding disorder or esophageal varices.
* Active parasitic infection or suspicion of an active parasitic infection, which, in the opinion of the site-Investigator, has not been previously evaluated or treated. Subjects presenting with signs of active parasitic infection or suspicion of active parasitic infection as assessed by current diarrhea and/or blood or mucus in stool will be referred to their clinical physician for further testing to rule out parasitic infection.
* Any other active infections judged at the discretion of the site-Investigator.
* Any other medical or psychological condition that, in the opinion of the site-investigator, may present an unreasonable risk to the study patient as a result of his/her participation in this clinical trial, may make patient's participation unreliable, or may interfere with study assessments. The specific justification for patients excluded under this criterion will be noted in study documents.
* Patient or his/her immediate family is a member of the investigational team.
* Pregnancy or breastfeeding.
* Women of children bearing potential who are not on highly-effective contraception.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan S Dellon, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - MNGI Digestive Health, P.A., Minneapolis, Minnesota
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dellon ES, Peterson KA, Mitlyng BL, Iuga A, Bookhout CE, Cortright LM, Walker KB, Gee TS, McGee SJ, Cameron BA, Galanko JA, Woosley JT, Eluri S, Moist SE, Hirano I. Mepolizumab for treatment of adolescents and adults with eosinophilic oesophagitis: a multicentre, randomised, double-blind, placebo-controlled clinical trial. Gut. 2023 Oct;72(10):1828-1837. doi: 10.1136/gutjnl-2023-330337. Epub 2023 Jul 9. PMID 37423717

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Followed by Mepolizumab 100 mg: Subjects will receive placebo subcutaneously (SQ) monthly for 3 months, followed by Mepolizumab 100 mg subcutaneously (SQ) monthly for 3 months. Mepolizumab will be administered with 2 SQ injections of placebo and 1 SQ injection of Mepolizumab 100 mg to maintain blinding.
  Mepolizumab 100 mg: Mepolizumab 100 mg subcutaneous injection
  Placebo: Saline subcutaneous injection
Period: Overall Study
Arm/Group | Mepolizumab 300 mg | Placebo, Followed by Mepolizumab 100 mg
Started | 32 | 34
Received Intervention | 32 | 33
Completed Month 3 | 31 | 33
Subsequent 3 Months of Treatment (Part 2) | 28 | 28
Completed Month 6 | 28 | 28
Completed | 27 | 26
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mepolizumab 300 mg | Placebo, Followed by Mepolizumab 100 mg | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 34 | 66
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (12) | 33.1 (9.8) | 35.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 21 | 18 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 31 | 33 | 64
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 30 | 33 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Dysphagia Score
Description: Dysphagia will be assessed by the Eosinophilic Esophagitis Symptom Activity Index (EEsAI) which measures dysphagia frequency, dysphagia severity, and food avoidance/modification behaviors. EEsAI scores range from 0 to 100, with higher scores indicating more severe symptoms. A decrease of ≥ 20 points is felt to be a meaningful clinical response and scores ≤ 20 representing clinical remission.
Time Frame: Baseline, Month 3 Post-Treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mepolizumab 300 mg | Placebo, Followed by Mepolizumab 100 mg
Number analyzed (Participants) | 31 | 33
score on a scale | 15.4 (18.1) | 8.3 (18)
Statistical Analysis 1: Comparison: Mepolizumab 300 mg vs Placebo, Followed by Mepolizumab 100 mg; Test type: Superiority; p = 0.14, ANCOVA

2. Secondary Outcome: Percent of Participants With a Clinical Remission (EEsAI Score of ≤ 20 Points)
Description: The EEsAI measures dysphagia frequency, dysphagia severity, and food avoidance/modification behaviors. EEsAI scores range from 0 to 100, with higher scores indicating more severe symptoms. A decrease of ≥ 20 points is felt to be a meaningful clinical response and scores ≤ 20 representing clinical remission.
Time Frame: After 3 months of treatment
Measure: Number; unit: percent of participants
Arm/Group | Mepolizumab 300 mg | Placebo, Followed by Mepolizumab 100 mg
Number analyzed (Participants) | 31 | 33
percent of participants | 6.45 | 6.06
Statistical Analysis 1: Comparison: Mepolizumab 300 mg vs Placebo, Followed by Mepolizumab 100 mg; Test type: Superiority; p = 0.95, Chi-squared

3. Secondary Outcome: Percent of Participants With a Clinical Response (EEsAI Score Decrease of ≥ 20 Points)
Description: as for outcome 2
Time Frame: After 3 months of treatment
Measure: Number; unit: percent of participants
Arm/Group | Mepolizumab 300 mg | Placebo, Followed by Mepolizumab 100 mg
Number analyzed (Participants) | 31 | 33
percent of participants | 35.48 | 21.21
Statistical Analysis 1: Comparison: Mepolizumab 300 mg vs Placebo, Followed by Mepolizumab 100 mg; Test type: Superiority; p = 0.20, Chi-squared

4. Secondary Outcome: Absolute Peak Eosinophil Count
Description: Absolute peak eosinophil (EOS) count (measured in EOS/hpf) after 3 months of treatment.
Time Frame: After 3 months of treatment
Measure: Mean (Standard Deviation); unit: eosinophils per high power field
Arm/Group | Mepolizumab 300 mg | Placebo, Followed by Mepolizumab 100 mg
Number analyzed (Participants) | 31 | 33
eosinophils per high power field | 35.7 (43) | 163 (133.1)
Statistical Analysis 1: Comparison: Mepolizumab 300 mg vs Placebo, Followed by Mepolizumab 100 mg; Test type: Superiority; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Number of Participants With Histologic Response as Assessed by Eosinophils Per High Powered Field
Description: Number of participants with a histologic response as assessed by having <15, ≤ 6, and ≤ 1 Eosinophils per high powered field (EOS/hpf).
Time Frame: After 3 months of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 300 mg | Placebo, Followed by Mepolizumab 100 mg
Number analyzed (Participants) | 31 | 33
Participants
  <15 eos/hpf | 13 | 1
  ≤6 eos/hpf | 7 | 1
  ≤1 eos/hpf | 3 | 1
Statistical Analysis 1: Comparison: Mepolizumab 300 mg vs Placebo, Followed by Mepolizumab 100 mg; <15 eos/hpf; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 2: Comparison: Mepolizumab 300 mg vs Placebo, Followed by Mepolizumab 100 mg; ≤6 eos/hpf; Test type: Superiority; p = 0.02, Chi-squared
Statistical Analysis 3: Comparison: Mepolizumab 300 mg vs Placebo, Followed by Mepolizumab 100 mg; ≤1 eos/hpf; Test type: Superiority; p = 0.27, Chi-squared

6. Secondary Outcome: Mean Change in Eosinophilic Esophagitis Endoscopic Reference Score (EREFS)
Description: Mean change in severity of endoscopic findings as measured by the EoE (Eosinophilic Esophagitis) Endoscopic Reference Score (EREFS). The EREFS, measures features of EoE including esophageal edema, rings, exudate, furrows, and strictures. The instrument grades edema as absent (0) or present (1); furrows as absent (0), mild (1), or severe (2); rings as absent (0), mild (1, subtle circumferential ridges), moderate (2, distinct rings) and severe (3, rings that impair passage of a standard adult diagnostic endoscope); exudates as absent (0), mild (1, less than 10% of the esophageal surface area) or severe (2, greater or equal to 10% of the esophageal surface area); and strictures as absent (0) or present (1) with an estimation of the minimal luminal diameter. Higher scores indicate more severe disease (range 0 - 9).
Time Frame: Baseline, 3 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mepolizumab 300 mg | Placebo, Followed by Mepolizumab 100 mg
Number analyzed (Participants) | 31 | 33
score on a scale | 1 (1.1) | 0.4 (1.3)
Statistical Analysis 1: Comparison: Mepolizumab 300 mg vs Placebo, Followed by Mepolizumab 100 mg; Test type: Superiority; p = 0.03, ANCOVA

7. Secondary Outcome: Mean Change in the Straumann Dysphagia Instrument (SDI) Score
Description: The Straumann Dysphagia Instrument (SDI) is a direct measure of dysphagia frequency and severity which is completed by participants and reported over the previous week. The score ranges from 0-9, with higher scores indicating more severe dysphagia.
Time Frame: Baseline, 3 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mepolizumab 300 mg | Placebo, Followed by Mepolizumab 100 mg
Number analyzed (Participants) | 31 | 33
score on a scale | 2.4 (1.7) | 2.7 (2.2)
Statistical Analysis 1: Comparison: Mepolizumab 300 mg vs Placebo, Followed by Mepolizumab 100 mg; Test type: Superiority; p = 0.44, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline through Month 6 post treatment assessments
Description: Adverse events were captured from time of consent (prior to group assignment) through Month 6.
Groups:
- Mepolizumab 300 mg: Baseline to Month 3: Subjects received Mepolizumab 300 mg subcutaneously (SQ) monthly for 3 months.
  Mepolizumab 300 mg subcutaneous injection
- Placebo Only to Month 3: Subjects received placebo subcutaneously (SQ) monthly for 3 months.
  Placebo: Saline subcutaneous injection
- Mepolizumab 300 mg Continuing to 6 Months: Subjects continued to receive Mepolizumab 300 mg subcutaneously (SQ) monthly through month 6.
  Mepolizumab 300 mg subcutaneous injection
- Placebo Switch to Mepolizumab 100 mg: Month 3 to Month 6: After the first 3 months of placebo, subjects received 3 months of Mepolizumab 100 mg subcutaneously (SQ) monthly. Mepolizumab was administered with 2 SQ injections of placebo and 1 SQ injection of Mepolizumab 100 mg to maintain blinding.
  Mepolizumab 100 mg subcutaneous injection
  Placebo: Saline subcutaneous injection
Arm/Group | Mepolizumab 300 mg: Baseline to Month 3 | Placebo Only to Month 3 | Mepolizumab 300 mg Continuing to 6 Months | Placebo Switch to Mepolizumab 100 mg: Month 3 to Month 6
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/34 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/32 | 0/34 | 2/28 | 0/28
Other Adverse Events (participants affected / at risk) | 13/32 | 19/34 | 12/28 | 18/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 300 mg: Baseline to Month 3 (N=32) | Placebo Only to Month 3 (N=34) | Mepolizumab 300 mg Continuing to 6 Months (N=28) | Placebo Switch to Mepolizumab 100 mg: Month 3 to Month 6 (N=28)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal decompression surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pre-existing lumbar degenerative disc disease requiring surgery
Orthopoedic Surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Left wrist surgery for arthritis
Corrective Jaw Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 300 mg: Baseline to Month 3 (N=32) | Placebo Only to Month 3 (N=34) | Mepolizumab 300 mg Continuing to 6 Months (N=28) | Placebo Switch to Mepolizumab 100 mg: Month 3 to Month 6 (N=28)
Injection site reaction (General disorders) | 9 (14) | 4 (4) | 8 (12) | 5 (5)
Injection site bruise (General disorders) | 1 (2) | 3 (4) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 3 (4) | 0 (0) | 3 (4)
COVID-19 (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (3) | 1 (1) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Sore Throat (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Esophageal Pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) — Pain in the esophagus
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) — Vomiting
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — Dysphagia
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) — Sinusitis
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) — Upper respiratory infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT03656380/Prot_SAP_000.pdf